CLINICAL TRIAL: NCT04192851
Title: Evaluation of "Tent-Pole" Grafting Technique for Reconstruction of Mandibular Ridge Vertical Defects (Clinical and Radiographic Study)
Brief Title: Evaluation of "Tent-Pole" Grafting Technique for Reconstruction of Mandibular Ridge Vertical Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Instructor of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tent-pole graft
Record Dates: First submitted 2019-12-07; First posted 2019-12-10 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Jaw Deformity
MeSH Terms: conditions — Jaw Abnormalities

STUDY DESIGN:
Intervention Model Description: This is a single-arm trial of 12 patients with mandibular large vertical defects treated using synthetic bone graft around titanium screws to tent out the soft tissue matrix.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tent Pole Grafting Technique (Experimental): * Bone graft [NanoBone® granulate 0,6 mm (24% Silica / 76% Hydroxylapatite)] is mixed with the patient blood and placed to cover the screws completely, the defect is overcorrected with particulate material in anticipation of future graft resorption.
  * PRF membrane is prepared by:
  Ten milliliters of whole venous blood will be collected in sterile glass test tubes without anticoagulant. Then the test tubes will be placed in a table centrifuge machine at 3000 revolutions per minute (rpm) for 10 minutes.After separation of PRF, the membrane is prepared compression device.
  Interventions: Procedure: Tent Pole Technique

INTERVENTIONS:
Procedure: Tent Pole Technique — * All patients were operated under local or general anaesthesia according to the case and patient tolerability.
  * The oral cavity was prepared by 0.12% chlorhexidine mouthrinses solution* for thirty seconds.
  * Full thickness incision down to the bone with blade no.15.
  * A periosteal elevator was used to perform mucoperiosteal flap.
  * Gentle elevation of the flap
  * Fixation of the screws over the alveolar ridge with about 5 mm of the screw threads will be exposed
  * Bone graft was mixed with the patient blood and placed to cover the screws completely.
  * PRF membrane was be placed over the grafted sites.
  * Repositioning of the flap and suturing with 3/0 black silk suture material

SUMMARY:
The aim of this study is to evaluate clinically and radio-graphically the efficiency of "Tent- Pole "grafting technique for reconstruction of anterior or posterior mandibular ridge defects using synthetic bone graft and Platelet Rich Fibrin (PRF) membrane.

DETAILED DESCRIPTION:
Various techniques have been described for the reconstruction of large vertical defects before implant placement . In this study we assessed the efficacy of tenting the periosteum and soft tissue matrix with titanium screws maintaining a space for the graft material in order to augment large vertical defects of mandibular ridge (anterior or posterior region) using data from 12 patients . After 6 months we assessed the increase in bone height and density.

ELIGIBILITY:
Inclusion Criteria:

* Patients with missing lower tooth or teeth and have a related large vertical bony defect .
* Patients with about 7mm residual bone hight and requiring about 5 mm increase in the vertical height of the mandibular alveolar ridge for future prosthetic rehabilitation.
* Patients with an acceptable oral hygiene and willing to improve it

Exclusion Criteria:

* Presence of infection or local lesions.
* Parafunctional habits.
* Current chemotherapy or radiotherapy.
* Heavy smokers.
* Alcohol or drug abuse.
* Medically compromised patients with diseases that affect passively the clinical procedure or result.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Pain assessment using Visual Analogue Scale | 2 weeks
  Pain was assessed through on a 10-point Visual Analogue Scale (VAS). (0-1= None, 2-4= Mild, 5-7= Moderate, 8-10= Severe)
Postoperative edema | 2 weeks
  Edema was evaluated by its ability to pit.The examiner fingers pressed into dependent area of the patient skin for 5 seconds. The finger sinks into the tissue and leave an impression when they are removed. The pitting was graded on a scale of +1 to +4 as follows:
  * 1 (trace) slight indentation rapid return to normal.
  * 2 (mild) the indentation returns to normal in a few seconds.
  * 3 (moderate) 6 mm indentation rebounds in 10-20 seconds.
  * 4 (severe) 8 mm indentation rebounds in more than 30 seconds.
Radiographic Evaluation for Bone Density using Cone Beam CT | 6 months
  A Cone Beam Computerized Tomography was obtained to assess the gained bone height &density.

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa M Abd ElFattah, BDS, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Abd El Aziz F Khalil, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Lydia N.F Melek, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Jensen SS, Terheyden H. Bone augmentation procedures in localized defects in the alveolar ridge: clinical results with different bone grafts and bone-substitute materials. Int J Oral Maxillofac Implants. 2009;24 Suppl:218-36. PMID 19885447
- [Background] Chiapasco M, Casentini P, Zaniboni M. Bone augmentation procedures in implant dentistry. Int J Oral Maxillofac Implants. 2009;24 Suppl:237-59. PMID 19885448
- [Background] Aghaloo TL, Moy PK. Which hard tissue augmentation techniques are the most successful in furnishing bony support for implant placement? Int J Oral Maxillofac Implants. 2007;22 Suppl:49-70. PMID 18437791
- [Background] Le B, Burstein J, Sedghizadeh PP. Cortical tenting grafting technique in the severely atrophic alveolar ridge for implant site preparation. Implant Dent. 2008 Mar;17(1):40-50. doi: 10.1097/ID.0b013e318166d503. PMID 18332757